CLINICAL TRIAL: NCT03150381
Title: Promoting Weight-Loss in African American Cancer Survivors in the Deep South
Acronym: DSNCARES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Monica L Baskin, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: X120329018
Record Dates: First submitted 2017-05-10; First posted 2017-05-12 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Weight Loss; Cancer
MeSH Terms: conditions — Weight Loss; Neoplasms

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single Blind (Participant)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Weight Loss Only (Active Comparator): Group-based behavioral weight loss intervention designed to reach clinically significant weight loss (~5-10% of baseline weight).
  Interventions: Behavioral: Weight Loss Only
- Weight Loss Plus (Experimental): Group-based behavioral weight loss intervention designed to reach clinically significant weight loss (~5-10% of baseline weight) plus community-level strategies to support healthy weight. Strategies are based on CDC's recommended community strategies and are developed by local contractors. They include expanded farmers markets/gardens, improvement to walking trails, etc.
  Interventions: Behavioral: Weight Loss Plus
- Control (Active Comparator): Educational materials and optional participation in community-wide cancer awareness activities.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Weight Loss Only — 24- month weight loss program (year 1: weekly in person meetings for 6 months, followed by 2 meetings per month for 3 months, then monthly for 3 months; year 2: monthly phone calls)
  Arms: Weight Loss Only
Behavioral: Weight Loss Plus — Participants will attend in-person weekly sessions (about 1.5 hours each) for 6 months and then twice a month for 3 months and monthly for 3 months. Sessions focus on behavioral techniques supporting healthy diet (including calorie restriction for weight loss) and achieving recommended amounts of physical activity per week. During 1-year weight loss maintenance, participants receive monthly motivational phone calls.
  Arms: Weight Loss Plus
Behavioral: Control — Participants receive quarterly newsletters containing generic cancer prevention messages and participate in community-wide cancer awareness educational sessions.
  Arms: Control

SUMMARY:
This study tests evidence-based strategies for weight loss among overweight and obesity cancer survivors and family members in rural Alabama.

DETAILED DESCRIPTION:
This is a 3-arm cluster randomized controlled study that compares a trained lay provided weight loss program vs. the same program plus community-based weight management strategies vs. general cancer prevention education on weight loss and other clinical outcomes (primary outcomes) and healthy behaviors, and psychosocial functioning (secondary outcomes).

ELIGIBILITY:
Inclusion Criteria:

* African American breast, colon, or prostate cancer survivor (Index Participant)
* Family member (support person) of African American breast, colon, or prostate cancer survivor (Family Member Participant)
* Live, work, or attend school in target county
* BMI >= 25 kg/m2

Exclusion Criteria:

* Pregnant or planning to become pregnant in the next year
* Known major medical or psychological condition known to influence body weight
* Uncontrolled hypertension (BP > 160 mmHg systolic or >100 mmHg diastolic)
* medicated or poorly controlled diabetes (glucose > 126) Cardiovascular event in the preceding 12 months
* History of gastric bypass or bariatric surgery
* History of psychiatric hospitalization in past 2 years
* History of substance abuse or eating disorder
* Any other condition by which a medical professional has suggested diet modification, physical activity and/or weight reduction would be contraindicated

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Weight | Baseline to 6 months
  Measured weight (nearest kg)

SECONDARY OUTCOMES:
Waist Circumference | Baseline to 24 months
  Measured circumference (nearest cm)
Lipids | Baseline to 24 months
  Measured total cholesterol, triglycerides, HDL, LDL, ratio (mg/dL)
Blood Pressure | Baseline to 24 months
  Measured blood pressure (mmHG) - systolic and diastolic
Weight | Baseline to 12 months
  Measured weight (nearest kg)
Weight | Baseline to 24 months
  Measured weight (nearest kg)
Social Support for Diet and Exercise Behaviors | Baseline to 6 months
  self report measure of social support (family, friend) in performing diet and exercise behaviors
Social Support for Diet and Exercise Behaviors | Baseline to 12 months
  self report measure of social support (family, friend) in performing diet and exercise behaviors
Social Support for Diet and Exercise Behaviors | Baseline to 24 months
  self report measure of social support (family, friend) in performing diet and exercise behaviors
Self Efficacy for Diet and Exercise Behaviors | Baseline to 6 months
  self report measure of confidence in performing diet and exercise behaviors
Self Efficacy for Diet and Exercise Behaviors | Baseline to 12 months
  self report measure of confidence in performing diet and exercise behaviors
Self Efficacy for Diet and Exercise Behaviors | Baseline to 24 months
  self report measure of confidence in performing diet and exercise behaviors
Automated Self-Administered 24-Hour Dietary Assessment Tool (ASA24) | Baseline to 6 months
  self report measure of dietary intake
Automated Self-Administered 24-Hour Dietary Assessment Tool (ASA24) | Baseline to 12 months
  self report measure of dietary intake
Automated Self-Administered 24-Hour Dietary Assessment Tool (ASA24) | Baseline to 24 months
  self report measure of dietary intake

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No